CLINICAL TRIAL: NCT03705949
Title: Impact of 0.1% Sodium Hyaluronate and 0.2% Sodium Hyaluronate on Postoperative Discomfort Following Cataract Extraction Surgery, a Comparative Study
Brief Title: Impact of 0.1% and 0.2% Sodium Hyaluronate on Postoperative Discomfort Following Phacoemulsification Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Collaborators: Naval Hospital, Athens (Other); George Papanicolaou Hospital (Other); Athinaiki General Clinic (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Associate Professor of Ophthalmology, Democritus University of Thrace
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 226/15-03-2018
Record Dates: First submitted 2018-10-11; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Active Comparator): Sodium Hyaluronate 0.1% drops
  Interventions: Drug: Sodium Hyaluronate 0.2% drops
- Control group (Active Comparator): Sodium Hyaluronate 0.2% drops
  Interventions: Drug: Sodium Hyaluronate 0.1% drops

INTERVENTIONS:
Drug: Sodium Hyaluronate 0.1% drops — Patients will be administered Drops of Sodium Hyaluronate 0.1% quid
  Other Names: Sodium Hyaluronate 0.1% drops (artificial tear medication)
  Arms: Control group
Drug: Sodium Hyaluronate 0.2% drops — Patients will be administered Drops of Sodium Hyaluronate 0.2% quid
  Other Names: Sodium Hyaluronate 0.2% drops (artificial tear medication)
  Arms: Study group

SUMMARY:
Primary objective of the study is the assessment of the patients' discomfort following cataract extraction surgery by means of phacoemulsification and intraocular lens implantation.

DETAILED DESCRIPTION:
Participants will be recruited from the Cataract Service of the University Hospital of Alexandroupolis (UHA), the Naval Hospital in Athens, the Papanikolaou General Hospital in Thessaloniki, and Athinaiki General Clinic in Athens in a consecutive-if-eligible basis. By means of a custom computer randomization program all participants will randomly populate either study group [who will receive fixed combination of tobramycin and dexamethasone (FCTD), (Tobradex, Alcon, Greece) quid for 3 weeks and 0.2 % sodium hyaluronate (Hylogel, Pharmex, Greece) quid for 6 weeks], and control group [who will receive Tobradex quid for 3 weeks and 0.1 % sodium hyaluronate (Hylocomod) quid for 6 weeks].

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of senile cataract with stage 2 or 3 nuclear opalescence according to the - Lens Opacities Classification System III (LOCS-3) grading scale

Exclusion Criteria:

1. Diagnosis or evidence of dry-eye-disease (DED)
2. IOP-lowering medications
3. Former incisional surgery
4. Former diagnosis of corneal disease
5. Diabetes
6. Autoimmune diseases
7. Mental diseases

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Surface Discomfort Index | 6 weeks
  A subjective parameter that quantifies corneal discomfort

SECONDARY OUTCOMES:
Break up time | 6 weeks
  An objective parameter that quantifies stability of tear film
Central Corneal Sensitivity | 6 weeks
  An objective parameter that quantifies corneal sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD, PhD, Study Director — University Hospital of Alexandroupolis, Democritus University of Thrace
Locations (1):
- University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

REFERENCES:
- [Derived] Ntonti P, Panagiotopoulou EK, Karastatiras G, Breyannis N, Tsironi S, Labiris G. Impact of 0.1% sodium hyaluronate and 0.2% sodium hyaluronate artificial tears on postoperative discomfort following cataract extraction surgery: a comparative study. Eye Vis (Lond). 2019 Feb 11;6:6. doi: 10.1186/s40662-019-0131-8. eCollection 2019. PMID 30805405